CLINICAL TRIAL: NCT07021014
Title: Improving Cardiovascular Health in Women With PTSD by Treating Trauma-Related Nightmares With NightWare
Brief Title: NightWare and Cardiovascular Health in Women With PTSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Ludeman Family Center for Women's Health Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-1948
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Post Traumatic Stress Disorder; Cardiovascular Diseases; Autonomic Dysfunction; Vascular Stiffness; Nightmare; Endothelial Dysfunction; Kidney Diseases; Renal Dysfunction; Trauma and Stressor Related Disorders
Keywords: Sleep; Trauma and Stressor Related Disorders; Post Traumatic Stress Disorder; Cardiovascular Diseases; Kidney Diseases; Renal Dysfunction; Autonomic Dysfunction
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Cardiovascular Diseases; Primary Dysautonomias; Kidney Diseases; Renal Insufficiency; Trauma and Stressor Related Disorders

STUDY DESIGN:
Intervention Model Description: Observational study (women with PTSD-related nightmares vs control group without PTSD-related nightmares); In women with PTSD-related nightmares only: randomized, double-blind, placebo (i.e., sham intervention) controlled parallel pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Experimental NightWare (Experimental): In women with PTSD-related nightmares randomized to the active condition, when the stress index is reached during sleep, NightWare will intervene with varying degrees of vibratory stimulation to the watch over a variable length of time to arouse the person out of the nightmare without awakening.
  Interventions: Device: NightWare
- Sham NightWare (Sham Comparator): In women with PTSD-related nightmares randomized to the sham condition, the NightWare intervention will not be enabled
  Interventions: Device: Sham NightWare
- Control Women without PTSD-related Nightmares (No Intervention): Age-matched women without PTSD-related nightmares will complete baseline testing only (no intervention).

INTERVENTIONS:
Device: NightWare — A wearable digital therapeutic platform consisting of an Apple Watch and iPhone pre-provisioned with Nightware intervention app that will deliver a mild vibration to the watch after detecting individual having a nightmare based on Nightware proprietary algorithm, arousing the individual and disrupting nightmare without awakening.
  Arms: Experimental NightWare
Device: Sham NightWare — NightWare decive will not deliver an intervention (i.e., no vibration)
  Arms: Sham NightWare

SUMMARY:
The purpose of this study is to determine whether NightWare therapeutic intervention improves biomarkers of vascular and renal function in premenopausal women with PTSD-related nightmares, and examine whether these improvements restore them to levels observed in age-matched women without PTSD.

DETAILED DESCRIPTION:
Women are disproportionally affected by posttraumatic stress disorder (PTSD), a debilitating mental health disorder that profoundly increases cardiovascular disease (CVD) risk. Biological processes including vascular dysfunction (i.e., impaired endothelial function, arterial stiffening), increased renin-angiotensin-aldosterone system (RAAS) activity, and altered renal vascular control and function may contribute to the pathophysiological link between PTSD and CVD. Sleep is a key regulator of cellular and tissue repair, free radical detoxification, oxidative stress, inflammation, autonomic and endocrine balance and crucial for cardiovascular health. Sleep disturbances due to nightmares are a hallmark symptom of PTSD that cause significant distress and may independently contribute to elevated CVD risk in individuals with PTSD. As such, interventions aimed at treating trauma-related nightmares are a promising therapeutic approach in ameliorating the cardiovascular consequences of PTSD.

NightWare™, a smart-watch based application that uses biometric data and vibrotactile feedback to disrupt nightmares, is an FDA approved digital therapeutic system for the treatment of nightmares in adults (≥22 years) with PTSD. While a preliminary study demonstrated that 30 days of NightWare treatment improved subjective sleep quality in Veterans, the influence of NightWare treatment on vascular and renal function in young women with PTSD-related nightmares is unknown. These investigations are critical among women who, despite having 2x greater prevalence of PTSD compared to men, and a differential progression of PTSD, CVD, and chronic kidney disease (CKD), are underrepresented in the literature.

Accordingly, the investigators will examine if the NightWare digital therapeutic system improves vascular and renal function in premenopausal women with PTSD-related nightmares, and whether these improvements restore them to levels observed in age-matched women without PTSD. We will employ 1) cross-sectional comparisons between two groups of women: those with PTSD and nightmares (PTSD group) and those without PTSD and nightmares (age-matched control group); and 2) a short-term (8-week) NightWare or sham intervention in women with nightmares related to PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by medical history
* Group Specific Eligibility
* PTSD Group
* Lifetime PTSD: screened using Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) and confirmed via Clinician Administered PTSD Scale for DSM-5 (CAPS-5)
* Prior trauma exposure: screened using Brief Trauma Questionnaire (BTQ)
* Self-report having repetitive nightmares contributing to disrupted sleep
* Poor overall sleep quality: PSQI score 6 or higher
* Control Group
* No lifetime PTSD: screened using PC-PTSD-5
* No prior trauma exposure: screened using BTQ
* Do not self-report having repetitive nightmares contributing to disturbed sleep

Exclusion Criteria:

* Pre-existing (e.g., diabetes, liver, kidney disease) or unstable medical condition (e.g., uncontrolled hypertension or active CVD or cancer) or systemic illness that would interfere with interpretation of the study outcomes
* Body Mass Index ≥ 40 kg/m2
* Use of medications that might influence cardiovascular or renal function (i.e., antihypertensive, lipid lowering medications, GLP-1/GIP RAs)
* Active infection (note, anyone with an active infection would become eligible once the infection has ended)
* Abnormal thyroid, liver, or kidney function testing during the screening examination or bloodwork. Abnormal kidney function defined as creatinine >1.3mg/dL. Abnormal liver function tests within 1.5x ULN. UCH Clinical Lab ULN for AST and ALT are 39 and 52, respectively. Women with TSH levels outside of the normal range (0.5-5.0 mLU/L) will be referred to their PCP and will be allowed study entry once their TSH levels are normalized > 3 months
* Plasma glucose >126 mg/dl under fasting conditions
* Use of insulin or sulfonylureas
* Pregnant, within 12 months postpartum or currently breast feeding
* Current history of substance (excluding marijuana) or alcohol abuse per the SCID-5. Adults with past substance or alcohol use disorders will be allowed to participate.
* Report elevated acute risk for suicidal self-directed violence warranting immediate hospitalization (e.g., suicidal ideation with intent, evaluated by the C-SSRS).
* Shift workers
* Diagnosis of active disorder of arousal from non-rapid eye movement sleep, rapid eye movement sleep behavior disorder, or narcolepsy
* Nocturia that causes awakening from sleep
* Epworth Sleepiness Scale: Question #8 score above "0" will prompt an additional question: Do you drive ("get behind the wheel") when you are drowsy? The answer must be "No" to be enrolled in the study due to safety concerns
* Known sleep walking or acting out dreams (contraindication to NightWare use)
* Diagnosis or suspicion of dementia
* Participants experiencing severe cognitive impairment or current psychiatric symptoms of such severity that would preclude participation (e.g., active psychosis, imminently suicidal)
* Current use of vitamin/supplements (including melatonin) or anti-inflammatory medications, participants will be included if they are willing to stop taking vitamin/supplements or anti-inflammatory medications 2 weeks prior to the first vascular visit.
* Current or planned participation in an interventional study during the present study
* Participants must have access to wireless internet and two power outlets where they sleep

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — cisgender premenopausal women
Enrollment: 36 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation (FMD) | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  FMD of the brachial artery, calculated as a percentage, is an index of vascular function. A higher number is a general indicator of better vascular function.

SECONDARY OUTCOMES:
Large artery elastic stiffness | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  Carotid-femoral pulse wave velocity (PWV). A higher number is a general indicator of worse vascular function.

OTHER OUTCOMES:
Large artery elastic stiffness-carotid artery | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  Carotid artery compliance using carotid artery ultrasound; a higher carotid artery compliance is a general indicator of better vascular function.
Autonomic function-baroreflex sensitivity | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  Cardiovagal baroreflex sensitivity (cBRS) measured using beat-to-beat time series of systolic blood pressures (finger photo-plethysmography) and R-R interval (three-lead electrocardiogram) will be recorded simultaneously at 1,000 Hz.
Autonomic function- heart rate variability | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  Heart rate variability
Blood pressure | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  Seated blood pressure measured in mmHg
Estimated glomerular filtration rate (eGFR) | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  Serum cystatin C, alongside demographic information, will be used to estimate kidney filtration of waste and excess water. A low eGFR can indicate renal dysfunction.
Renal vascular control | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  Peak change in renal vascular resistance in response to sympathoexcitation via cold pressor test
Renal functional reserve | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  Peak change in creatinine clearance (calculated using urine creatinine, serum creatinine, urine flow rate) following ingestion of oral protein
Pittsburgh Sleep Quality Index (PSQI) | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  Sleep questionnaire with a scale of 0 to 21 with a higher score indicating a significant sleep disturbance
Pittsburgh Sleep Quality Index Addendum for PTSD (PSQI-A) | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  Sleep questionnaire to assess frequency of seven disruptive nocturnal behaviors; scores range from 0-21 with higher scores indicating more severe PTSD-related sleep disturbances.
PTSD Checklist for DSM-5 (PCL-5) | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  Presence and severity of PTSD symptoms questionnaire; scores range from 0-80 with higher scores indicating more severe PTSD symptoms.
Nightmare Disorder Index (NDI) | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  5-item questionnaire related to nightmares; scores range from 0-20 with higher score indicates more severe nightmare symptoms.
Columbia Suicide Severity Rating Scale (CSSR-S) | PTSD vs controls at baseline. In PTSD group only, change with NightWare vs Sham (measured before and after 8 weeks of NightWare or sham conditions).
  Questionnaire used for suicide risk assessment; categorizes level of suicide risk (low, moderate, high) based on responses to questions about suicidal ideation and behavior.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado CCTSI CTRC, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No